CLINICAL TRIAL: NCT00177775
Title: Whey Protein Concentrate 40% (WPC-40) Made of Milk of Immunized Cows to Aid in the Prevention of Relapse of Clostridium Difficile-Diarrhea: A Prospective, Randomized, Controlled Phase II Study - Version 5.1.B
Brief Title: Whey Protein Concentrate 40% Made of Milk of Immunized Cows to Aid in the Prevention of Relapse of Clostridium Difficile-Diarrhea
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study is completed and analysis completed
Sponsor: University of Pittsburgh (Other)
Collaborators: MucoVax, BV, the Netherlands (Unknown)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB# 0412033
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Positive C-Diff Culture

INTERVENTIONS:
Drug: MucoMilk product

SUMMARY:
The primary objective of this study is to assess the safety of the investigational agent, MucoMilk®, a polyclonal-antibody enriched Whey Protein Concentrate 40% (WPC-40) made of milk of immunized cows. Secondary objectives will investigate the effectiveness of MucoMilk® as an aid in the prevention of relapse of C. difficile-associated diarrhea (CDAD).

DETAILED DESCRIPTION:
This is a single-center, prospective, controlled, randomized, open-label study. Sixty subjects will be randomized 2:1 to receive MucoMilk® (n=40) or to the control arm with no specific product intervention (n=20). There is no effective FDA-approved treatment to prevent recurrence of CDAD that is being withheld from subjects who will be randomized to the control arm.

The sponsor will prepare sequentially numbered batches of MucoMilk® for the entire 2-week dosing period, or 42 packets, and will prepare a randomization table that will be held in confidence by the University of Pittsburgh Investigational Drug Service (IDS) pharmacist. Each subject will be assigned a sequential study number (i.e. 1, 2, 3, etc.) as they are enrolled in the study. Upon enrollment, research staff will contact the IDS pharmacist to obtain the subject's study number and randomization assignment (MucoMilk® or no specific product intervention). Research staff will not have access to the randomization table.

Subjects assigned to receive MucoMilk® will be given a box containing 14 leaflets numbered "Day 1" to "Day 14". Each leaflet consists of 3 packets labeled "morning", "noon", and "evening" connected by perforated paper. Subjects will be provided with one box and instructed not to alter their diet during the two-week course.

At the University of Pittsburgh, it is anticipated that up to 150 subjects will need to be screened in order to enter 60 subjects on study. Subjects may participate in this study for up to 63 days.

Subjects will be managed and followed per institutional infection control guidelines for C. difficile containment regardless of assigned study group. Subjects will receive appropriate treatment for comorbid conditions based on the judgement of the treating physician and practice guidelines. With the exception of investigational agents, any clinically indicated concomitant medications for symptomatic relief or support will be allowed upon recommendation and approval of the investigator.

For this trial, the safety of MucoMilk® will be determined by passive self-reporting in a subject diary and active surveillance by preset interview of any adverse events. In addition, a physical exam and extensive hematologic and biochemical testing will be performed before and after MucoMilk® administration.

Efficacy will be examined by assessing CDAD relapse rates. A relapse of CDAD will be reached when, in comparison with the day before, stools have become looser and either (1) the frequency of stools has increased for 2 consecutive days, or (2) on a single day the frequency increases by > 3 stools, or (3) occurrence of > 6 stools/day on any day. In this respect, CDAD relapse will be defined as "probable" if occurring as described for the first 18 days following MucoMilk® initiation with a negative C. diff toxin assay or "proven" if occurring at any time with a positive C. diff toxin assay. A subject will be considered a treatment failure if s/he meets the above criteria for a CDAD relapse.

Subjects who cannot or will not be included in this study will be asked to be followed for 60 days off-study for any adverse reaction(s) or CDAD relapses per subject diary documentation. These subjects may receive treatment for CDAD outside of this study as standard of care but will not be offered any study product or intervention through randomization.

3.3 Clinical and Laboratory Evaluations: Subjects may be either inpatients or outpatients during their participation in this study. Inpatient study visits will take place at UPMC Presbyterian, UPMC Montefiore, or UPMC Shadyside. Outpatient study visits will take place at the Infectious Disease Clinic in the Falk Medical Building. Each study visit will last about one hour depending on the procedures to be done at that visit.

All procedures performed in this study are research-required with the exception of the antibiotic treatment for CDAD initiated at the Diagnosis Visit and any stool toxin assays performed to confirm suspected CDAD relapse as these are both standard of care for CDAD. The investigator will review the results of all evaluations, and these results will become part of the subject's research record.

It may be necessary for the subject to make additional visit(s) during participation in this study to have any of the study procedures listed below repeated in the event of unforeseen or unanticipated abnormal results; difficulties in sample shipping, processing, or testing; and/or if the subject experiences any changes in his/her physical condition.

Screening Procedures:

Screening Visit for all subjects will occur within 3 days prior to Day 1 or will be combined with the Day 1 Visit as subjects may be randomized if currently receiving or have completed standard antibiotic therapy for CDAD. Subjects will be asked to read and sign the informed consent before any study procedures are performed. Evaluations to be done at this visit include:

* Complete physical examination.
* Collection of demographic data, medication history, chronic health score, and primary/relapse CDAD episode information.
* Female subjects of childbearing potential will be given a urine pregnancy test, which must be negative.

Subjects currently on a standard antibiotic course for CDAD with oral/intravenous metronidazole and/or vancomycin will continue this therapy for a minimum of 10 days per standard of care at the discretion of the study physician.

Experimental Procedures:

Day 1 Visit will occur during or within 3 days after Screening. If diarrhea has recurred and CDAD relapse is suspected, stool sample for toxin assay by ELISA/cell test, culture, and microscopy. If positive for CDAD, the subject will be taken off study and followed as per standard of care for CDAD relapse. Evaluations include:

* Karnofsky and EORTC GI scores.
* 45ml blood draw for hematology (Hgb, WBC w/diff, platelets), renal function (creatinine, urea, electrolytes), liver function (ALT, AST, alkaline phosphatase, albumin, glucose, total protein, bilirubin), lipids, IgE, and for storage.
* Female subjects of childbearing potential will be given a urine pregnancy test, which must be negative.
* Distribution of subject diary for recording of any adverse event(s) and the number and consistency of all stools.

At the completion of these evaluations, MucoMilk® subjects will receive enough study product for entire 14-day dosing period, be counseled on proper storage and administration by the study staff, and be given a study agent diary to record compliance.

Day 7 to 9 Visit will be conducted by telephone for outpatients or by visit for inpatients to review stool frequency and consistency and any perceived adverse events from MucoMilk®, if applicable. If a CDAD relapse is suspected based on this review, the subject will be asked to provide a stool sample for toxin assay. If positive for CDAD, the subject will be taken off MucoMilk® if applicable, off study, and followed as per standard of care for CDAD relapse.

Follow-Up Procedures:

Day 18 to 21 Visit evaluations include:

* Targeted physical exam.
* Karnofsky and EORTC GI scores.
* 45ml blood draw for hematology, renal and liver function tests, lipids, IgE, and for storage.
* If diarrhea has recurred and CDAD relapse is suspected, stool sample for toxin assay by ELISA/cell test, culture, and microscopy.
* Collection of any unused investigational product and study agent diary.
* Subject diary review. Subjects will continue to record any adverse event(s) and the number and consistency of all stools during the follow-up period.

Through Day 60 weekly visits will be conducted by telephone or visit to review bowel movements and stool consistency. If a CDAD relapse is suspected based on any review, the subject will be asked to provide a stool sample for toxin assay. If positive for CDAD, the subject will be taken off study and followed as per standard of care for CDAD relapse. The occurrence and time to the occurrence of any new relapse in this period will be evaluated as well. Subjects who complete the study through Day 60 with no relapse of CDAD will be asked to return their diary, discharged from study participation, and referred back to their primary care physician for follow-up.

3.4 Storage of Biological Samples: During this study, serum samples collected on Day 1 and on Day 18 to 21 will be labeled with the subject's study identification number and date collected; processed; frozen; and stored at MucoVax for future testing that is part of this study, including investigation of antibodies directed against C. difficile and its toxins. Also, the presence of human antibodies directed against bovine immunoglobulins may be examined. The sponsor will have sole control over these samples, which will be stored for an indefinite period of time. Subjects will not be notified of the results of these future studies as the information collected will not apply to the management of their disease at the time these tests are done. If these samples are provided to secondary investigators, these samples, devoid of all subject identifiers and rendered anonymous, will be obtained from the sponsor by the secondary investigator. The secondary investigator will not have direct access to any subject identifiers or related subject information.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects must meet all of the following inclusion criteria:

* Willingness and ability to comply with all study requirements, to fully understand all elements of informed consent, and to provide written informed consent.
* Confirmed CDAD by ELISA toxin assay or cell test.
* Are currently receiving or have received standard antibiotic treatment for CDAD with oral/intravenous metronidazole and/or vancomycin for a minimum of 10 days per standard of care at the discretion of the study physician.
* Resolution of diarrhea to a maximum of 3 stools per day following completion of antibiotic therapy.
* Ability to tolerate fluids by mouth or by feeding tube.
* Have passage of stools.

Exclusion Criteria:

Subjects will not be eligible to participate in this study if any of the following exclusion criteria apply:

* Unable to provide informed consent.
* History of lactose intolerance.
* Cannot tolerate fluids by mouth or by feeding tube, or are judged by the attending physician unfit to receive fluids by mouth or by feeding tube.
* Have received an investigational drug within 4 weeks prior to study entry.
* Have underlying gastrointestinal tract disease characterized by diarrhea or unformed stools.
* Are currently receiving any antidiarrheal medications.
* Current use of an ileostomy or colostomy.
* History of milk allergy.
* Current use of Saccharomyces boulardii, Lactinex, or Culturelle preparations at start of study. (S. boulardii is a non-colonizing yeast species purported to support gastrointestinal tract function. It has been widely studied and used to help prevent post-antibiotic diarrhea.)
* Reside outside of the United States.
* Cannot speak or read English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-04; Study Completion 2005-08

PRIMARY OUTCOMES:
To investigate the effectiveness of MucoMilk®

SECONDARY OUTCOMES:
To assess the safety of MucoMilk

CONTACTS AND LOCATIONS:
Overall Officials: Peter Veldkamp, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States